CLINICAL TRIAL: NCT00090233
Title: Safety and Efficacy of Pentavalent (G1, G2, G3, G4 , and P1) Human-Bovine Reassortant Rotavirus Vaccine in Healthy Infants
Brief Title: Rotavirus Efficacy and Safety Trial (REST)(V260-006)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: V260-006; 2004_012
Record Dates: First submitted 2004-08-25; First posted 2004-08-27 (Estimated); Results first posted 2011-05-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-09

CONDITIONS: Rotavirus Infections
MeSH Terms: conditions — Rotavirus Infections | interventions — RotaTeq; Rotavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): RotaTeq
  Interventions: Biological: Rotateq™
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Comparator: Placebo

INTERVENTIONS:
Biological: Rotateq™ — 3 doses of 2.0 mL RotaTeq administered orally. Dose 1 will be given at study entry, Dose 2 will be given 4-10 weeks after Dose 1, Dose 3 will be given 4-10 weeks after Dose 2.
  Other Names: V260
  Arms: 1
Biological: Comparator: Placebo — 3 doses of 2.0 mL Placebo to RotaTeq administered orally. Dose 1 will be given at study entry, Dose 2 will be given 4-10 weeks after Dose 1, Dose 3 will be given 4-10 weeks after Dose 2.
  Arms: 2

SUMMARY:
This study was designed to evaluate the safety of the investigational rotavirus vaccine and the efficacy to prevent rotavirus gastroenteritis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants

Exclusion Criteria:

* None Specified

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 69274 (Actual)
Dates: Start 2001-01; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Vesikari T, Matson DO, Dennehy P, Van Damme P, Santosham M, Rodriguez Z, Dallas MJ, Heyse JF, Goveia MG, Black SB, Shinefield HR, Christie CD, Ylitalo S, Itzler RF, Coia ML, Onorato MT, Adeyi BA, Marshall GS, Gothefors L, Campens D, Karvonen A, Watt JP, O'Brien KL, DiNubile MJ, Clark HF, Boslego JW, Offit PA, Heaton PM; Rotavirus Efficacy and Safety Trial (REST) Study Team. Safety and efficacy of a pentavalent human-bovine (WC3) reassortant rotavirus vaccine. N Engl J Med. 2006 Jan 5;354(1):23-33. doi: 10.1056/NEJMoa052664. PMID 16394299
- [Derived] Itzler R, Koch G, Matson DO, Gothefors L, Van Damme P, Dinubile MJ, Heaton PM. Robustness of the healthcare utilization results from the Rotavirus Efficacy and Safety Trial (REST) evaluating the human-bovine (WC3) reassortant pentavalent rotavirus vaccine (RV5). BMC Pediatr. 2010 Jun 11;10:42. doi: 10.1186/1471-2431-10-42. PMID 20540778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 356 sites in Belgium, Costa Rica, Finland, Germany, Guatemala, Italy, Jamaica, Mexico, Puerto Rico, Sweden, Taiwan, and the United States from 12 Jan 2001 first patient in (FPI) to 06 Oct 2004 last patient in (LPI).
Pre-assignment Details: Participants with: history of congenital abdominal disorders, intussusception, or abdominal surgery; history of
  known prior rotavirus disease, chronic diarrhea, or failure to thrive were excluded from the trial before
  assignment to groups.
Groups:
- RotaTeq™: Three oral doses (~6.5x10^7 to ~1.2x10^8 IU/dose) of RotaTeq™ (rotavirus vaccine, live, oral, pentavalent) administered at 3 separate visits scheduled 4 to 10 weeks (28 to 70 days) apart with up to 42 days of safety follow-up after each vaccination, and follow-up for acute gastrointestinal episodes (AGEs) through the first rotavirus season postvaccination. The rotavirus season for each site was prospectively determined using historical epidemiologic data.
- Placebo: Placebo matching RotaTeq™ administered at 3 separate visits scheduled 4 to 10 weeks (28 to 70 days) apart with up to 42 days of safety follow-up after each vaccination, and follow-up for acute gastrointestinal episodes (AGEs) through the first rotavirus season postvaccination. The rotavirus season for each site was prospectively determined using historical epidemiologic data.
Period: Overall Study
Arm/Group | RotaTeq™ | Placebo
Started | 34644 (Evaluated by data safety monitoring board (DSMB) when they recommended stopping enrollment) | 34630 (Evaluated by data safety monitoring board when they recommended stopping enrollment)
Vaccinated at Visit 1 | 34035 (Randomized Not vaccinated 609) | 34003 (Randomized Not vaccinated 627)
Vaccinated at Visit 2 | 31052 | 31066
Vaccinated at Visit 3 | 29667 | 29598
Completed | 29645 (Does not include participants who discontinued prior to the 42 day safety follow-up) | 29565 (Does not include participants who discontinued prior to the 42 day safety follow-up)
Not Completed | 4999 | 5065
Not completed — Randomized Not Vaccinated (Visit 1) | 609 | 627
Not completed — Adverse Event | 214 | 198
Not completed — Lost to Follow-up | 68 | 95
Not completed — Protocol Violation | 960 | 1022
Not completed — Withdrawal by Subject | 182 | 211
Not completed — Moved | 203 | 189
Not completed — Other | 1211 | 1160
Not completed — Data not available at data cut-off point | 1552 | 1563

BASELINE CHARACTERISTICS:
Groups:
- RotaTeq™: Three oral doses (~6.5x10^7 to ~1.2x10^8 IU/dose) of RotaTeq™ (rotavirus vaccine, live, oral, pentavalent) administered at 3 separate visits scheduled 4 to 10 weeks (28 to 70 days) apart.
- Placebo: Placebo matching RotaTeq™ administered at 3 separate visits scheduled 4 to 10 weeks (28 to 70 days) apart.
- Total: Total of all reporting groups
Arm/Group | RotaTeq™ | Placebo | Total
Number analyzed (Participants) | 34644 | 34630 | 69274
Age, Customized [Number; unit: Participants] — The eligibility for this study was to enroll infants 6-12 weeks of age; however infants that were 5 weeks and under, and infants who were 12 weeks and over were inadvertently enrolled outside these ranges. Those infants who received at least 1 dose of study vaccine, were followed for safety.
  Participants
    5 Weeks of Age and Under | 1 | 4 | 5
    6 to 12 Weeks of Age | 34551 | 34527 | 69078
    Over 12 Weeks of Age | 92 | 99 | 191
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17058 | 17101 | 34159
  Male | 17586 | 17529 | 35115
Race/Ethnicity [Number; unit: participants]
  White | 23772 | 23788 | 47560
  Hispanic American | 4963 | 4911 | 9874
  Black | 2908 | 2941 | 5849
  Multi Racial | 1815 | 1817 | 3632
  Asian | 536 | 552 | 1088
  Native American | 531 | 514 | 1045
  Other | 119 | 107 | 226

OUTCOME MEASURES:

1. Primary Outcome: Intussusception Within 42 Days Following Any Dose of RotaTeq™/Placebo
Description: Number of participants with confirmed intussusception within 42 days after each vaccination with RotaTeq™/placebo.
Time Frame: Within 42 days following any dose of RotaTeq™/placebo
Population: All participants in the study were followed for potential cases of intussusception.
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 34002 | 33969
Participants | 6 | 5
Statistical Analysis 1: Comparison: RotaTeq™ vs Placebo; Test type: Non-Inferiority or Equivalence — Relative Risk ≤10.0 (non-inferiority margin); p = 0.006, Exact binomial test — p≤ 10/11, where p is proportion of participants with intussusception in vaccine group relative to total number of participants with intussusception. Based on conditional binomial approach. Adjusted for group-sequential design; Exact binomial test adjusted for group-sequential design; relative risk = 1.6, 95% CI [0.4 to 6.4]

2. Secondary Outcome: G1 Serum Neutralizing Antibody (SNA) Responses Against Rotavirus
Description: Number of participants with a 3-fold rise or greater in G1 Serum neutralizing antibody (SNA) responses against rotavirus from baseline to postdose 3.
Time Frame: 14 days following the 3rd vaccination
Population: Per Protocol Population among participants in Finland using Per-Protocol Case Definition
Measure: Number; unit: Participants
Groups:
- RotaTeq™: Participants randomized to treatment with RotaTeq™ tested with data available for analysis excluding protocol violators, participants with invalid data based on laboratory determinations, participants with wildtype rotavirus detected in the stool, or with samples taken outside the range of 9 to 33 days postdose 3.
- Placebo: Participants randomized to treatment with Placebo tested with data available for analysis excluding protocol violators, participants with invalid data based on laboratory determinations, participants with wildtype rotavirus detected in the stool, or with samples taken outside the range of 9 to 33 days postdose 3.
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 117 | 89
Participants | 95 | 8
Statistical Analysis 1: Comparison: RotaTeq™; Test type: Superiority or Other; p < 0.001, Exact binomial test — p≥42%, where p is proportion of participants with ≥3-fold rise in antibody titer from Predose 1 to Postdose 3 in vaccine group. Based on binomial approach; Proportion = 81.2, 95% CI [72.9 to 87.8]

3. Primary Outcome: Occurrence of Rotavirus Disease Caused by Serotypes G1, G2, G3 and G4 That Occurs 14 Days Following the 3rd Vaccination
Description: Rotavirus gastroenteritis cases consist of all participants with one or more episodes classified as positive. Multiple positive episodes for one participant are counted as a single case.
Time Frame: At least 14 days following the 3rd vaccination through the first full rotavirus season
Population: Per Protocol Population Using Per-Protocol Case Definition
Measure: Number; unit: Participants
Groups:
- RotaTeq™: The number of participants randomized to treatment with RotaTeq™ is different from the number analyzed because some participants were excluded due to protocol violations and/or participants without follow-up and/or participants classified as unevaluable due to detection of wildtype rotavirus in the stool prior to 14 days Postdose 3; incomplete clinical and/or laboratory results; or stool samples collected out of day range.
- Placebo: The number of participants randomized to treatment with Placebo is different from the number analyzed because some participants were excluded due to protocol violations and/or participants without follow-up and/or participants classified as unevaluable due to detection of wildtype rotavirus in the stool prior to 14 days Postdose 3; incomplete clinical and/or laboratory results; or stool samples collected out of day range.
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 2207 | 2305
Participants | 82 | 315
Statistical Analysis 1: Comparison: RotaTeq™ vs Placebo; Test type: Superiority or Other; p < 0.001, Exact binomial test — Efficacy≥35%. Based on p≤.65/(.65+k), where p is proportion of participants with outcome in vaccine group relative to total number of participants with outcome, k is ratio of follow-up time; placebo/vaccine. Based on conditional binomial approach; Exact binomial test; Efficacy=1-Relative Risk = 74.0, 95% CI [66.8 to 79.9] — Efficacy = 1-RR, expressed as a percentage; the RR is the incidence in the vaccine group / the incidence in the placebo group

4. Secondary Outcome: Occurrence of Hospital Admissions and Visits to Emergency Departments (or the Equivalent at International Sites) for Rotavirus Disease Associated With Serotypes G1, G2, G3, or G4
Description: Health Outcomes Substudy - Occurrence of hospital admissions and emergency department visits for episode(s) of rotavirus gastroenteritis associated with serotypes G1, G2, G3, or G4 by treatment group. Occurrence was expressed as the annual number of events per 1000 person-years.
Time Frame: At least 14 days following the 3rd vaccination
Population: Per Protocol Population Using Per-Protocol Case Definition
Measure: Number; unit: Annual # of events per 1000 person-years
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 28646 | 28488
Annual # of events per 1000 person-years
  Hospital admissions | 6 | 144
  Emergency department visits | 14 | 213
Statistical Analysis 1: Comparison: RotaTeq™ vs Placebo; Test type: Superiority or Other; p < 0.001, Poisson regression — Rate Reduction>0%; Poisson regression with generalized estimating equations. Validated with Van Elteren's extension of Wilcoxon Rank Sum test; Risk Ratio (RR) = 94.5, 95% CI [91.2 to 96.6] — Risk ratio of rate of hospitalizations and emergency department visits between treatment groups. Reported here are results after 12 additional emergency department visits were identified among placebo recipients and data were re-analyzed

5. Secondary Outcome: Efficacy of a 3-dose Regimen of RotaTeq™ Against Moderate-to-severe Rotavirus Disease (Clinical Score >8) Caused by Serotypes G1, G2, G3, and G4 Occurring at Least 14 Days Following the Third Dose.
Description: Number of participants with rotavirus gastroenteritis whose clinical score was >8 for the first episode and for the worst episode. Scores evaluated the intensity and duration of diarrhea, vomiting, fever, and behavioral symptoms. The total score for an episode is equal to the sum of the scores for each of the symptoms [range: total score 0 (best) to 24 (worst)].
Time Frame: At least 14 days following the 3rd vaccination through the first rotavirus season
Population: Per Protocol Population Using Per-Protocol Case Definition
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 2201 | 2292
Participants
  First episode scores | 48 | 262
  Worst episode scores | 49 | 265
Statistical Analysis 1: Comparison: RotaTeq™ vs Placebo; Test type: Superiority or Other; p < 0.001, Exact binomial test — Efficacy>0%. Based on p< 1/(1+k), where p is proportion of participants with outcome in vaccine group relative to total number of participants with outcome, and k is ratio of follow-up time; placebo / vaccine. Based on conditional binomial approach; Efficacy=1-Relative Risk = 81.5, 95% CI [74.9 to 86.7] — Estimated value is based on the worst episode scores

6. Secondary Outcome: Efficacy of a 3-dose Regimen of RotaTeq™ Against Severe Rotavirus Disease (Clinical Score > 16) Caused by Serotypes G1, G2, G3, and G4 Occurring at Least 14 Days Following the Third Dose
Description: Number of participants with rotavirus gastroenteritis whose clinical score was >16 for the first episode and for the worst episode. Scores evaluated the intensity and duration of diarrhea, vomiting, fever, and behavioral symptoms. The total score for an episode is equal to the sum of the scores for each of the symptoms [range: total score 0 (best) to 24 (worst)].
Time Frame: At least 14 days following the 3rd vaccination through the first rotavirus season
Population: Per Protocol Population Using Per-Protocol Case Definition
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 2198 | 2271
Participants
  First episode scores | 1 | 51
  Worst episode scores | 1 | 51
Statistical Analysis 1: Comparison: RotaTeq™ vs Placebo; Test type: Superiority or Other; p < 0.001, Exact binomial test — Efficacy>0%. Based on p< 1/(1+k), where p is proportion of participants with outcome in vaccine group relative to total number of participants with outcome, and k is ratio of follow-up time; placebo/vaccine. Based on conditional binomial approach; Efficacy=1-Relative Risk = 98.0, 95% CI [88.3 to 100]

7. Secondary Outcome: Seroprotection/Seroconversion for Hepatitis B, Haemophilus Influenzae Type b, Diphtheria, Tetanus, & Polio Types 1,2,& 3 Who Received COMVAX™, INFANRIX™, IPOL™ & PREVNAR™ Concomitantly With RotaTeq™ Versus Placebo
Description: The number of participants who achieved seroprotection/seroconversion to hepatitis B, Haemophilus influenzae type b, diphtheria, tetanus, & polio types 1, 2, & 3, per established criteria.
Time Frame: 42 days following third dose
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 558 | 592
Participants
  Hepatitis B (N=202, N=214) | 197 | 203
  Haemophilus influenzae type b (N=558, N=592) | 417 | 426
  Diphtheria (N=136, N=144) | 136 | 142
  Tetanus (N=132, N=140) | 132 | 140
  Polio type 1 (N=341, N=360) | 328 | 349
  Polio type 2 (N=341, N=359) | 311 | 326
  Polio type 3 (N=341, N=359) | 324 | 343
Statistical Analysis 1: Comparison: RotaTeq™ vs Placebo; Test type: Non-Inferiority or Equivalence — Difference (vaccine-placebo) in seroprotection rates was greater than -.10 (non-inferiority margin); p < 0.001, Miettenen and Nurminen — p<0.001 was obtained for all comparisons. pv - pp ≥-.10, where p is proportion of participants who achieved seroprotection in the vaccine and placebo groups, respectively

8. Secondary Outcome: Geometric Mean Antibody Titer(s) (GMT) to Pertussis Toxin (PT), Pertussis Filamentous Haemagglutinin (FHA), and Pertussis Pertactin
Description: Measurement of immune response in the group that received RotaTeq™ and the group that received placebo was performed by determining geometric mean antibody titers to Pertussis Toxin (PT), Pertussis Filamentous Haemagglutinin (FHA), and Pertussis Pertactin. Antibody titers were measured with an indirect, non-competitive, enzyme immunoassay (EIA).
Time Frame: 42 days following third dose
Population: Per Protocol Population; excluding protocol violators and participants with invalid data based on laboratory determinations.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 59 | 78
ELISA units/mL
  Pertussis PT | 20.18 [17.10 to 23.81] | 22.73 [19.59 to 26.37]
  Pertussis FHA | 55.69 [48.01 to 64.59] | 64.33 [55.41 to 74.69]
  Pertussis Pertactin | 34.77 [26.46 to 45.70] | 59.17 [46.21 to 75.76]
Statistical Analysis 1: Comparison: RotaTeq™ vs Placebo; The GMT Ratio between RotaTeq™ and Placebo (GMTR) for Pertussis PT was used for analysis; Test type: Non-Inferiority or Equivalence — GMTR was greater than 0.5 (non-inferiority margin); p < 0.001, t-test, 1 sided; t-test on natural log of titers; GMTR for Pertussis PT = 0.9, 95% CI 2-sided [0.7 to 1.1]
Statistical Analysis 2: Comparison: RotaTeq™ vs Placebo; The GMT Ratio between RotaTeq™ and Placebo (GMTR) for Pertussis FHA was used for analysis; Test type: Non-Inferiority or Equivalence — GMTR was greater than 0.5 (non-inferiority margin); p < 0.001, t-test, 1 sided; t-test on natural log of titers; GMTR for Pertussis FHA = 0.9, 95% CI 2-sided [0.7 to 1.1]
Statistical Analysis 3: Comparison: RotaTeq™ vs Placebo; The GMT Ratio between RotaTeq™ and Placebo (GMTR) for Pertussis Pertactin was used for analysis; Test type: Non-Inferiority or Equivalence — GMTR was greater than 0.5 (non-inferiority margin); p = 0.193, t-test, 1 sided; t-test on natural log of titers; GMTR for Pertussis Pertactin = 0.6, 95% CI 2-sided [0.4 to 0.8]

9. Secondary Outcome: Geometric Mean Antibody Titer(s) (GMT) to Pneumococcal Serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F
Description: Measurement of immune response in the group that received RotaTeq™ and the group that received placebo was performed by determining geometric mean antibody titers to pneumococcal serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F. Serum antibody titers to type-specific pneumococcal polysaccharides were determined by an EIA.
Time Frame: 42 days following third dose
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms/mL
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 185 | 198
micrograms/mL
  Pneumococcal serotype 4 (N=181, N=196) | 1.13 [0.99 to 1.29] | 0.96 [0.84 to 1.09]
  Pneumococcal serotype 6B (N=185, N=198) | 2.39 [1.93 to 2.95] | 1.72 [1.38 to 2.13]
  Pneumococcal serotype 9V (N=166, N=181) | 1.90 [1.66 to 2.19] | 1.78 [1.55 to 2.04]
  Pneumococcal serotype 14 (N=178, N=198) | 4.24 [3.39 to 5.29] | 4.33 [3.55 to 5.28]
  Pneumococcal serotype 18C (N=166, N=180) | 2.60 [2.30 to 2.94] | 2.02 [1.76 to 2.32]
  Pneumococcal serotype 19F (N=180, N=196) | 1.97 [1.61 to 2.42] | 1.84 [1.55 to 2.20]
  Pneumococcal serotype 23F (N=185, N=198) | 1.71 [1.41 to 2.07] | 1.50 [1.24 to 1.80]
Statistical Analysis 1: Comparison: RotaTeq™ vs Placebo; The GMT Ratio between RotaTeq™ and Placebo (GMTR) for pneumococcal serotype 4 was used for analysis; Test type: Non-Inferiority or Equivalence — GMTR was greater than 0.5 (non-inferiority margin); p < 0.001, t-test, 1 sided; t-test on natural log of titers; GMTR for pneumococcal serotype 4 = 1.2, 95% CI [1.0 to 1.4]
Statistical Analysis 2: Comparison: RotaTeq™ vs Placebo; The GMT Ratio between RotaTeq™ and Placebo (GMTR) for pneumococcal serotype 6B was used for analysis; Test type: Non-Inferiority or Equivalence — GMTR was greater than 0.5 (non-inferiority margin); p < 0.001, t-test, 1 sided; t-test on natural log of titers; GMTR for pneumococcal serotype 6B = 1.4, 95% CI 2-sided [1.0 to 1.9]
Statistical Analysis 3: Comparison: RotaTeq™ vs Placebo; The GMT Ratio between RotaTeq™ and Placebo (GMTR) for pneumococcal serotype 9V was used for analysis; Test type: Non-Inferiority or Equivalence — GMTR was greater than 0.5 (non-inferiority margin); p < 0.001, t-test, 1 sided; t-test on natural log of titers; GMTR for pneumococcal serotype 9V = 1.1, 95% CI 2-sided [0.9 to 1.3]
Statistical Analysis 4: Comparison: RotaTeq™ vs Placebo; The GMT Ratio between RotaTeq™ and Placebo (GMTR) for pneumococcal serotype 14 was used for analysis; Test type: Non-Inferiority or Equivalence — GMTR was greater than 0.5 (non-inferiority margin); p < 0.001, t-test, 1 sided; t-test on natural log of titers; GMTR for pneumococcal serotype 14 = 1.0, 95% CI 2-sided [0.7 to 1.3]
Statistical Analysis 5: Comparison: RotaTeq™ vs Placebo; The GMT Ratio between RotaTeq™ and Placebo (GMTR) for pneumococcal serotype 18C was used for analysis; Test type: Non-Inferiority or Equivalence — GMTR was greater than 0.5 (non-inferiority margin); p < 0.001, t-test, 1 sided; t-test on natural log of titers; GMTR for pneumococcal serotype 18C = 1.3, 95% CI 2-sided [1.1 to 1.6]
Statistical Analysis 6: Comparison: RotaTeq™ vs Placebo; The GMT Ratio between RotaTeq™ and Placebo (GMTR) for pneumococcal serotype 19F was used for analysis; Test type: Non-Inferiority or Equivalence — GMTR was greater than 0.5 (non-inferiority margin); p < 0.001, t-test, 1 sided; t-test on natural log of titers; GMTR for pneumococcal serotype 19F = 1.1, 95% CI 2-sided [0.8 to 1.4]
Statistical Analysis 7: Comparison: RotaTeq™ vs Placebo; The GMT Ratio between RotaTeq™ and Placebo (GMTR) for pneumococcal serotype 23F was used for analysis; Test type: Non-Inferiority or Equivalence — GMTR was greater than 0.5 (non-inferiority margin); p < 0.001, t-test, 1 sided; t-test on natural log of titers; GMTR for pneumococcal serotype 23F = 1.1, 95% CI 2-sided [0.9 to 1.5]

ADVERSE EVENTS:
Time Frame: Participants in this study were followed for all serious adverse events (SAEs) and other adverse events (AEs), for up to 42 days following each study vaccination
Description: Participants listed in SAE tables (34904-RotaTeq; 34862-Placebo) are those who received study treatment. Other AEs were reported for a pre-defined subset who received ≥1 dose (4808-RotaTeq; 4796-Placebo). Although a participant may have had ≥ 2 AEs they are counted only once in a category. The same participant may appear in different categories.
Groups:
- RotaTeq™: Three oral doses (~6.5x10^7 to ~1.2x10^8 IU/dose) of RotaTeq™ (rotavirus vaccine, live, oral, pentavalent) administered at 3 separate visits scheduled 4 to 10 weeks (28 to 70 days) apart.
  The Not Completed total includes participants discontinued at any time before the completion of the third study vaccination and/or the 42-day safety follow-up period post vaccination 3.
- Placebo: Placebo matching RotaTeq™ administered at 3 separate visits scheduled 4 to 10 weeks (28 to 70 days) apart.
  The Not Completed total includes participants discontinued at any time before the completion of the third study vaccination and/or the 42-day safety follow-up period post vaccination 3.
Arm/Group | RotaTeq™ | Placebo
Serious Adverse Events (participants affected / at risk) | 863/34904 | 955/34862
Other Adverse Events (participants affected / at risk) | 4000/4800 | 4047/4787
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ (N=34904) | Placebo (N=34862)
Anaemia (Blood and lymphatic system disorders) | 7 | 3
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 2 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cyanosis (Cardiac disorders) | 3 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 1
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 1
Coarctation of the aorta (Congenital, familial and genetic disorders) | 0 | 2
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 1
Congenital intestinal malformation (Congenital, familial and genetic disorders) | 1 | 1
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1
Cystic fibrosis (Congenital, familial and genetic disorders) | 1 | 1
Developmental glaucoma (Congenital, familial and genetic disorders) | 0 | 1
Glycogen storage disease type ib (Congenital, familial and genetic disorders) | 1 | 0
Hip dysplasia (Congenital, familial and genetic disorders) | 2 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Kidney malformation (Congenital, familial and genetic disorders) | 1 | 0
Polycystic liver disease (Congenital, familial and genetic disorders) | 0 | 1
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 2
Retinoblastoma (Congenital, familial and genetic disorders) | 0 | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 | 2
Chalazion (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Anal fissure (Gastrointestinal disorders) | 3 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 2
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anal skin tags (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 7 | 6
Diarrhoea (Gastrointestinal disorders) | 9 | 21
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 2 | 4
Faecaloma (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 29 | 17
Haematemesis (Gastrointestinal disorders) | 3 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 3
Infantile colic (Gastrointestinal disorders) | 2 | 2
Inguinal hernia (Gastrointestinal disorders) | 11 | 8
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 1
Intussusception (Gastrointestinal disorders) | 13 | 22
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 1
Regurgitation of food (Gastrointestinal disorders) | 1 | 2
Retching (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Volvulus of bowel (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 23 | 20
Brain death (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Death (General disorders) | 1 | 4
Drowning (General disorders) | 0 | 1
Fever neonatal (General disorders) | 2 | 1
Hernia (General disorders) | 1 | 0
Injection site inflammation (General disorders) | 1 | 0
Irritability (General disorders) | 9 | 4
Near sudden infant death syndrome (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 43 | 49
Sudden death (General disorders) | 1 | 0
Sudden infant death syndrome (General disorders) | 7 | 9
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Milk allergy (Immune system disorders) | 4 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess neck (Infections and infestations) | 1 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1
Adenovirus infection (Infections and infestations) | 1 | 0
Amoebic dysentery (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 2 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Botulism (Infections and infestations) | 2 | 0
Bronchiolitis (Infections and infestations) | 215 | 253
Bronchitis (Infections and infestations) | 25 | 20
Bronchitis acute (Infections and infestations) | 3 | 3
Bronchitis acute viral (Infections and infestations) | 0 | 1
Bronchitis chronic (Infections and infestations) | 1 | 2
Bronchitis viral (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 11 | 6
Campylobacter intestinal infection (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 6
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Chest wall abscess (Infections and infestations) | 1 | 0
Clostridium colitis (Infections and infestations) | 0 | 1
Coxsackie viral infection (Infections and infestations) | 0 | 1
Croup infectious (Infections and infestations) | 8 | 5
Cystitis (Infections and infestations) | 2 | 0
Dysentery (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 3 | 2
Eczema infected (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Enterovirus infection (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 2
Exanthema subitum (Infections and infestations) | 3 | 2
Febrile infection (Infections and infestations) | 2 | 3
Gastroenteritis (Infections and infestations) | 73 | 127
Gastroenteritis adenovirus (Infections and infestations) | 4 | 1
Gastroenteritis rotavirus (Infections and infestations) | 3 | 18
Gastroenteritis salmonella (Infections and infestations) | 2 | 4
Gastroenteritis viral (Infections and infestations) | 8 | 6
Gastrointestinal infection (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
Haemophilus sepsis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 5 | 6
Kawasaki's disease (Infections and infestations) | 5 | 0
Laryngitis (Infections and infestations) | 12 | 6
Laryngotracheitis (Infections and infestations) | 2 | 0
Laryngotracheo bronchitis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 7 | 4
Lower respiratory tract infection (Infections and infestations) | 0 | 3
Meningitis (Infections and infestations) | 4 | 2
Meningitis aseptic (Infections and infestations) | 2 | 2
Meningitis bacterial (Infections and infestations) | 1 | 1
Meningitis enteroviral (Infections and infestations) | 0 | 1
Meningitis haemophilus (Infections and infestations) | 0 | 1
Meningitis streptococcal (Infections and infestations) | 2 | 0
Meningitis viral (Infections and infestations) | 3 | 4
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 4 | 1
Otitis externa (Infections and infestations) | 2 | 0
Otitis media (Infections and infestations) | 28 | 24
Otitis media acute (Infections and infestations) | 3 | 2
Parainfluenzae virus infection (Infections and infestations) | 2 | 0
Parotitis (Infections and infestations) | 1 | 0
Perianal abscess (Infections and infestations) | 2 | 0
Perineal abscess (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 2 | 2
Pertussis (Infections and infestations) | 6 | 7
Pharyngitis (Infections and infestations) | 2 | 3
Pneumococcal bacteraemia (Infections and infestations) | 1 | 0
Pneumococcal infection (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 55 | 58
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 1 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 5 | 2
Pneumonia viral (Infections and infestations) | 1 | 3
Pseudocroup (Infections and infestations) | 0 | 2
Pyelocystitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 22 | 27
Pyelonephritis acute (Infections and infestations) | 16 | 12
Respiratory syncytial virus infection (Infections and infestations) | 10 | 6
Respiratory tract infection (Infections and infestations) | 13 | 14
Respiratory tract infection viral (Infections and infestations) | 3 | 2
Rhinitis (Infections and infestations) | 1 | 1
Roseola (Infections and infestations) | 2 | 1
Salmonellosis (Infections and infestations) | 0 | 2
Scrotal infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 7 | 4
Septic shock (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Tonsillitis streptococcal (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 2 | 0
Tuberculosis of peripheral lymph nodes (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 27 | 15
Urinary tract infection (Infections and infestations) | 38 | 29
Urosepsis (Infections and infestations) | 0 | 6
Varicella (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 14 | 17
Viral pharyngitis (Infections and infestations) | 0 | 1
Viral rash (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 4
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 3 | 6
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 5
Femur fracture (Injury, poisoning and procedural complications) | 1 | 5
Fractured skull depressed (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 3 | 2
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2
Injury asphyxiation (Injury, poisoning and procedural complications) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 3 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 4 | 2
Skull fracture (Injury, poisoning and procedural complications) | 7 | 7
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 4
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Body temperature increased (Investigations) | 1 | 0
Occult blood positive (Investigations) | 6 | 3
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 4
Cow's milk intolerance (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 19 | 23
Diet refusal (Metabolism and nutrition disorders) | 5 | 4
Failure to thrive (Metabolism and nutrition disorders) | 2 | 4
Feeding disorder (Metabolism and nutrition disorders) | 2 | 0
Feeding disorder neonatal (Metabolism and nutrition disorders) | 0 | 1
Food intolerance (Metabolism and nutrition disorders) | 0 | 2
Hyperinsulinaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 2
Weight gain poor (Metabolism and nutrition disorders) | 1 | 2
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 | 0
Growth retardation (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Pineal parenchymal neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anoxic encephalopathy (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 17 | 9
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 4 | 2
Febrile convulsion (Nervous system disorders) | 6 | 4
Hemiplegia (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 2
Hypotonia (Nervous system disorders) | 1 | 0
Hypoxic encephalopathy (Nervous system disorders) | 1 | 1
Infantile spasms (Nervous system disorders) | 1 | 3
Intraneural cyst (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 3
Spinal cord haemorrhage (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Apathy (Psychiatric disorders) | 0 | 1
Breath holding (Psychiatric disorders) | 2 | 0
Crying (Psychiatric disorders) | 5 | 5
Eating disorder (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 1
Staring (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 1
Balanitis (Reproductive system and breast disorders) | 1 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 1
Phimosis (Reproductive system and breast disorders) | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 | 11
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial hyperactivity (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neonatal apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 | 5
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2
Urticaria pigmentosa (Skin and subcutaneous tissue disorders) | 0 | 1
Child abuse (Social circumstances) | 1 | 1
Child neglect (Social circumstances) | 0 | 1
Overfeeding of infant (Social circumstances) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 2
Haemorrhage (Vascular disorders) | 0 | 1
Pallor (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ (N=4800) | Placebo (N=4787)
Conjunctivitis (Eye disorders) | 315 | 339
Abdominal pain upper (Gastrointestinal disorders) | 53 | 40
Constipation (Gastrointestinal disorders) | 188 | 214
Diarrhoea (Gastrointestinal disorders) | 1047 | 1022
Flatulence (Gastrointestinal disorders) | 273 | 282
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 62 | 59
Infantile colic (Gastrointestinal disorders) | 70 | 65
Regurgitation of food (Gastrointestinal disorders) | 175 | 183
Teething (Gastrointestinal disorders) | 196 | 165
Vomiting (Gastrointestinal disorders) | 613 | 644
Injection site pain (General disorders) | 216 | 228
Irritability (General disorders) | 881 | 862
Pyrexia (General disorders) | 1970 | 2056
Bronchiolitis (Infections and infestations) | 200 | 185
Bronchitis (Infections and infestations) | 79 | 73
Candida nappy rash (Infections and infestations) | 46 | 51
Ear infection (Infections and infestations) | 94 | 107
Gastroenteritis (Infections and infestations) | 447 | 454
Influenza (Infections and infestations) | 89 | 72
Nasopharyngitis (Infections and infestations) | 276 | 277
Oral candidiasis (Infections and infestations) | 185 | 188
Otitis media (Infections and infestations) | 624 | 602
Pharyngitis (Infections and infestations) | 60 | 57
Respiratory tract infection (Infections and infestations) | 97 | 83
Rhinitis (Infections and infestations) | 348 | 337
Upper respiratory tract infection (Infections and infestations) | 1230 | 1279
Viral infection (Infections and infestations) | 105 | 121
Decreased appetite (Metabolism and nutrition disorders) | 68 | 67
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45 | 46
Agitation (Psychiatric disorders) | 215 | 180
Crying (Psychiatric disorders) | 160 | 190
Restlessness (Psychiatric disorders) | 63 | 69
Cough (Respiratory, thoracic and mediastinal disorders) | 471 | 456
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 293 | 294
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 222 | 254
Wheezing (Respiratory, thoracic and mediastinal disorders) | 52 | 51
Dermatitis (Skin and subcutaneous tissue disorders) | 47 | 25
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 106 | 120
Eczema (Skin and subcutaneous tissue disorders) | 129 | 110
Rash (Skin and subcutaneous tissue disorders) | 167 | 153

LIMITATIONS AND CAVEATS:
70,301 participants randomized, 69,274 evaluated, when DSMB first recommended ending enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.